CLINICAL TRIAL: NCT06151756
Title: Video Mobile Applique Supported Teaching Used in Nursing Skill Training Effects on Students' Academic Success Problem Solving Critical Thinking Levels
Brief Title: Video Mobile Applique Supported Teaching Used in Nursing Skill Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sevil Şahin, Assoc Prof Dr, TC Erciyes University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019/03
Record Dates: First submitted 2023-11-14; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Nurse's Role
Keywords: Student nurse; Mobile applicability; Skills training; Problem solving; Critical thinking.

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial was designed. According to randomization in a computer environment of 200 students who meet the criteria for inclusion in the study, the intervention and control group were divided into two groups. This study was conducted in a university faculty of health sciences nursing department students with the aim of examining the impact of video mobile application-supported teaching utilized in nursing skills training on students' academic success, problem solving and critical thinking levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video mobile application supported education (Other): In order to ensure standardization in the expression of all skills, a video flow plan was prepared and recordings were conducted in accordance with this plan. The videos were organized in a way that the practitioner narrates all the steps of the procedure, with being visible and audible. Before the application, each video was watched repeatedly by the research team and necessary arrangements were performed. Then, the videos created about the applications were uploaded to the mobile application-based web system. After the systematic preparations were completed, trainings on the system and usage were provided to the instructors in charge of the skill practices. In addition, all students were trained on research, the system, and usage, and were provided with the opportunity to download the mobile application to their phones.
  Interventions: Behavioral: Video Supported Mobile Application
- Control (No Intervention): The students in the control group, on the other hand, were subjected to standardized training in the skills laboratory without watching any videos after the theoretical information provided in the course. While the students were practicing, they were evaluated by the relevant instructors according to the process steps in the "Basic Nursing Skills Learning Guide". In both groups, students were informed about the research and evaluated in terms of inclusion criteria. Prior to the start of the intervention, all students were asked to fill the student introduction form, the Problem Solving Inventory and the California Critical Thinking Disposition Scale.

INTERVENTIONS:
Behavioral: Video Supported Mobile Application — The video-supported mobile application was developed to be interactively utilized on smartphones. T
  Arms: Video mobile application supported education

SUMMARY:
This study was conducted in a university faculty of health sciences nursing department students with the aim of examining the impact of video mobile application-supported teaching utilized in nursing skills training on students' academic success, problem solving and critical thinking levels.A randomized controlled trial was designed.The study was conducted l with second-year students of the department of nursing at faculty of health sciences. The research was finalised with the participation of 167 students, 83 in the intervention group and 84 in the control group. Data were collected through Student Identification Form, Problem Solving Inventory, California Critical Thinking Disposition Scale and Basic Nursing Skills Learning Guide.

DETAILED DESCRIPTION:
Students in the intervention group were subjected to watch app videos via the mobile app before implementing skills. Students in the control group were subjected to standard training in the skills laboratory without watching any video after the theoretical knowledge described in the course. The data were collected through the Student demonstration form, the problem solving Inventory, the California critical thinking tendency scale and the Basic Nursing skills Learning Guide.

3.5. Data collection In line with the process steps in the Basic Nursing Skills Learning Guide, video recordings were carried out in the Nursing Skills Laboratory of our Faculty for each application in the Healthy Living and Nursing Module IX course. In order to ensure standardization in the expression of all skills, a video flow plan was prepared and recordings were conducted in accordance with this plan. The videos were organized in a way that the practitioner narrates all the steps of the procedure, with being visible and audible. Before the application, each video was watched repeatedly by the research team and necessary arrangements were performed. Then, the videos created about the applications were uploaded to the mobile application-based web system. After the systematic preparations were completed, trainings on the system and usage were provided to the instructors in charge of the skill practices. In addition, all students were trained on research, the system, and usage, and were provided with the opportunity to download the mobile application to their phones.

Initially, the theoretical parts of the skill practices within the scope of the Healthy Living and Nursing Module IX course were taught face-to-face in the course. Student rotation was established for the intervention in accordance with randomization. The practices of the students in the control group were carried out between 8.30-12.30 in the morning, while the practices of the intervention group were carried out between 13.30-17.30. While the students in the control group were practicing in the laboratory, the system was activated, the videos were made accessible to the students and only the students in the intervention group were allowed to watch the skill videos 3 times. The students in the intervention group participated in their own practices in the afternoon after watching the skill videos. The students in the control group, on the other hand, were subjected to standardized training in the skills laboratory without watching any videos after the theoretical information provided in the course. While the students were practicing, they were evaluated by the relevant instructors according to the process steps in the "Basic Nursing Skills Learning Guide".

In both groups, students were informed about the research and evaluated in terms of inclusion criteria. Prior to the start of the intervention, all students were asked to fill the student introduction form, the Problem Solving Inventory and the California Critical Thinking Disposition Scale. After the skill practices were finalized, all students were asked to fill the Problem Solving Inventory and California Critical Thinking Disposition Scale again. At the same time, after all the practices related to the course were completed, the students were examined and their academic achievement scores were evaluated after the application. After the applications were finished, the videos were made accessible to all students, including the students in the control group.

ELIGIBILITY:
Inclusion Criteria:

Students;

* Who were enrolled in the second year of the nursing department in the 2022-2023 academic year,
* Who attended the Healthy Living and Nursing Module IX course, Who participated in the respiratory system and gastrointestinal system practices in this course .
* Who agreed to participate in the study

Exclusion Criteria:

Students;

* Who did not attend the courses,
* Who worked as health care assistants,
* Who did not agree to participate in the study.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 167 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Problem Solving Inventory(PSI) | One mounth.
  PSI is a 6-point Likert-type scale consisting of 35 items ("I always act like this" 1 point, "I usually act like this" 2 points, "I frequently act like this" 3 points, "I sometimes act like this" 4 points, "I rarely act like this" 5 points, "I never act like this" 6 points). The scale has three sub-dimensions: "Confidence in problem solving ability", "Approach avoidance", and "Personal control". Items numbered 9, 22, 29 are excluded from the scoring. Items numbered 1, 2, 3, 4, 11, 13, 14, 15, 17, 21, 25, 26, 30 and 34 are reverse scored statements. The score range of the inventory is between 32-192 and the average score is 80. Values above the average indicate that the person is inadequate in problem solving, while values below the average indicate that the person is adequate in problem solving

CONTACTS AND LOCATIONS:
Overall Officials: Erciyes Universty, Study Director — Erciyes Üniversitesi Sağlık Bilimleri Fakültesi
Locations (1):
- Sevil Güler, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is nı plan